CLINICAL TRIAL: NCT02358447
Title: SPECT-CT for Assessment of Patients Before and After Navigated and Conventional Total Knee Arthroplasty.
Brief Title: SPECT-CT for Assessment of Total Knee Arthroplasty in Navigated and Non-navigated Total Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: Kantonsspital Baselland Bruderholz (Other)
Responsible Party: Principal Investigator, Michael Tobias Hirschmann, PD Dr. med., Kantonsspital Baselland Bruderholz
Other Study IDs: SPECT/CT-TKR_001_MH; 380/09 (Other: Ethikkommission beider Basel)
Record Dates: First submitted 2015-01-02; First posted 2015-02-09 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Osteoarthritis; X-rays; Effects
Keywords: total knee arthroplasty; total knee prothesis; Spectrometry, X-Ray Emission; SPECT/CT; measurement of TKA component position
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- SPECT/CT before/after navigated TKR: SPECT/CT in patients before and after navigated TKR (assessment of bone tracer uptake, 3D CT component position)
  Interventions: Procedure: TKR
- SPECT/CT before/after conventional TKR: SPECT/CT in patients before and after conventional TKR (assessment of bone tracer uptake, 3D CT component position)
  Interventions: Procedure: TKR

INTERVENTIONS:
Procedure: TKR — non-navigated versus computer-navigated total knee replacement

SUMMARY:
By the comparison of two operation methods navigated and non-navigated TKR with SPECT/CT we want to show wich method has the better outcome.

DETAILED DESCRIPTION:
With SPECT/CT we want to controll the clinical outcome of patients who underwent a navigated or a non-navigated TKR.

ELIGIBILITY:
Inclusion Criteria:

* Total Knee prosthesis (primary)
* >18 years

Exclusion Criteria:

* pregnancy
* lactating women
* endocrine diseases
* tumour diseases
* posttraumatic osteoarthritis of the knee
* previous infection of the knee
* medicaments which influence the metabolism of the bone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Paitents before and after total knee replacement surgery
Sampling Method: Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2010-04; Primary Completion 2017-07 (Actual); Study Completion 2018-10-23 (Actual)

PRIMARY OUTCOMES:
which operation method is the best in terms of outcome and SPECT/CT imaging | five years

SECONDARY OUTCOMES:
Improvement in the post-treatment | five years

CONTACTS AND LOCATIONS:
Overall Officials: MIchael T. Hirschmann, MD, Principal Investigator — Dept. of Orthop. Surgery and Traumatology, Kantonsspital Baselland - Bruderholz, Unitverstity of Basel, Switzerland
Locations (1):
- Kantonsspital Baselland, Bruderholz, Bruderholz, Basel-Landschaft, Switzerland